CLINICAL TRIAL: NCT00688480
Title: Do Xanthine Oxidase Inhibitors Reduce Both Left Ventricular Hypertrophy and Endothelial Dysfunction in Cardiovascular Patients With Renal Dysfunction?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A. D. Struthers (Other)
Responsible Party: Sponsor-Investigator, A. D. Struthers, Head Of Cardiovascular and Diabetes Medicine, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MK001
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Disease; Left Ventricular Hypertrophy
Keywords: CKD; LVH; Echo LVH; Chronic Stage 3
MeSH Terms: conditions — Kidney Diseases; Hypertrophy, Left Ventricular; Bronchiolitis Obliterans Syndrome | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Placebo Comparator): CKD Stage 3 (estimated GFR 30 - 60 ml/min/1.73m2), Echo LVH
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Placebo — 1 capsule, orally for 9 months
  Arms: I
Drug: Allopurinol — Allopurinol 300 mg once/day orally, 9 months
  Arms: 2

SUMMARY:
Cardiovascular related disease is the main cause of death in patients with kidney disease, and "oxidative stress" is thought to be a major contributor by promoting thickening of the heart muscle and stiffening of the arteries. Allopurinol, a drug used safely in the treatment of gout for many years, has been found to dramatically reduce "oxidative stress". It is therefore hoped that it also reduce the thickened heart muscle and stiffened arteries. If it did, it is likely to reduce the appallingly high cardiac death rate in this group of kidney disease patients.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3
* Echo LVH

Exclusion Criteria:

* Known heart failure
* Patients already on Allopurinol
* Patients with gout
* Patients with hepatic disease
* Contraindications to MRI, including severe claustrophobia
* Current immunosuppressive therapy, chlorpropamide, theophylline, 6- mercaptopurine
* Malignancy or other life threatening disease
* Pregnancy or lactating women
* Patients unable to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Primary objective is to see if Allopurinol reduces left ventricular hypertrophy (LVH) in this group of CKD patients | 9 months

SECONDARY OUTCOMES:
Secondary objective is to see if Allopurinol reduces endothelial dysfunction in this group of CKD patients | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan D Struthers, BSc, MD, FRCP, FESC, Principal Investigator — University of Dundee
Locations (1):
- Division of Medicine and Therapeutics, Ninewells Hospital & Medical School, Dundee, United Kingdom